CLINICAL TRIAL: NCT04660045
Title: A Phase II Trial of Early Intervention With Acalabrutinib in Patients With CLL at High Risk for Richter's Transformation
Brief Title: Early Intervention With Acalabrutinib in Patients With High Risk CLL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company supplying drug/funding ceased support.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-11022876
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Chronic Lymphocytic Leukemia; CLL/SLL
Keywords: CLL; untreated
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib (Experimental): Acalabrutinib 100 mg will be administered orally twice daily continuously in 28-day cycles until treatment is discontinued for any reason.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib, oral, 100 mg BID, continuous
  Other Names: CALQUENCE; ACP-196

SUMMARY:
This study evaluates the effectiveness of acalabrutinib treatment in patients with chronic lymphocytic leukemia (CLL) deemed at high risk for Richter's Transformation (RT). This is a single arm study. Enrolled patients will initiate therapy with acalabrutinib and will dose continuously. While on study, subjects will be monitored monthly for the first 3 months, then every three months thereafter until disease progression, discontinuation due to toxicity, death, or study completion.

DETAILED DESCRIPTION:
This is a multi-center, single arm, Phase II clinical trial to investigate the effectiveness of acalabrutinib treatment within 6 months of chronic lymphocytic leukemia (CLL) diagnosis for patients with CLL deemed at high risk for Richter's Transformation (RT).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.
* The time from diagnosis to consent should be ≤6 months.
* Subject must be ≥ 18 years of age.
* Subject must have diagnosis of CLL/SLL based upon 2018 iwCLL Guidelines.
* Rai stage 0-2 disease without indication for treatment as defined by the 2018 iwCLL guidelines
* Subject must have high risk CLL as defined by any one of the following:

  * NOTCH1 mutated (classic frameshift mutation only)
  * Unmutated V4-39 B cell receptor usage
  * Pathogenic c-MYC mutations
  * Complex karyotype, (by CpG/oligodeoxynucleotide stimulation)
  * Deletion 17p, or presence of TP53 mutation
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
* PT/PTT/INR within 1.5 x the ULN
* Adequate renal function defined by serum creatinine less than 2 x ULN
* Adequate hepatic function:

  * ALT/AST less than 2x ULN
  * Tbili less than 1.5 X ULN unless bilirubin elevation is due to Gilbert's syndrome (total bilirubin <3)
* Subject must have adequate bone marrow function.

  * Absolute neutrophil count ≥1.0 x103/μL
  * Hemoglobin ≥ 11.0 g/dL
  * Platelets ≥ 100 x 103/μL

Exclusion Criteria:

* Previous exposure to any systemic anti-cancer therapy as a treatment for CLL, including but not limited to chemotherapy, immunotherapy, radiotherapy, or investigational therapy. Note, patients treated with chemotherapy for a prior non-hematologic malignancy if more than 5 years earlier are eligible.
* Subject with a history of malignancy except for non-melanoma skin cancers. Subjects treated with curative intent via methods of local resection and or locally targeted anticancer treatment and are free of malignancy for at least 5 years from treatment end will be allowed to enroll.
* Subject requires chronic immunosuppressive therapy for any reason or was treated with immunosuppressive therapy within 6 months of study entry.
* Subjects with a history of autoimmune hemolytic anemia or immune thrombocytopenia purpura.
* Subject has prolymphocytic leukemia.
* Active bleeding, or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
* Subject requires warfarin or equivalent vitamin K antagonist
* Uncontrolled or active significant infection,
* History of or suspected or confirmed PML
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
* Patients with stroke or CNS hemorrhage within 6 months
* Pregnant or breastfeeding

  * Women of childbearing potential (WCBP) who are sexually active with heterosexual partners must agree to use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib.
* Major surgical procedure within 28 days of first dose of study drug. If a subject had surgery, they must have recovered adequately from any toxicity or complications before the first dose of study drug.
* Has difficulty with or is unable to swallow oral medication or has significant gastrointestinal disease that would limit absorption of oral medication.
* Subject is known to be positive for human immunodeficiency virus (HIV)
* Active hepatitis C, as confirmed by being positive for Hep C RNA by PCR
* Active hepatitis B infection documented by a positive PCR for Hep B DNA. If hepatitis B serology is positive for hepatitis B core antibody, but Hep B DNA PCR is negative, patient is eligible to enroll.
* Subject requires strong CYP 3A4/5 inhibitors or inducers (Appendix B).
* Subject requires proton pump inhibitors. (Subjects that can transition to an H2 antagonist are allowed to enroll.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who do not develop Richter's Transformation (RT) within 5 years of study drug administration | 5 years

SECONDARY OUTCOMES:
Event-free survival | 5 years
  Measured from time of study drug administration to time of progression, transformation to a more aggressive histology, treatment discontinuation due to toxicity, or death from any cause.
Progression-free survival | 5 years
  Measured from time of study drug administration to progression or death, measured in months.
Progression-free survival in patients with TP53 disruption | 5 years
  For subjects with TP53 disruption present at baseline, measured from time of study drug administration to progression or death, measured in months.
Overall survival | 5 years
  Measured from time of study drug administration to death from any cause, measured in months.
Percentage of subjects who do not develop Richter's Transformation within 2 years of study drug administration | 2 years
Median time to development of RT | 5 years
  Measured from time of study drug administration
Safety of early interventional acalabrutinib in patients with chronic lymphocytic leukemia (CLL) at high risk for Richter's Transformation | 5 years
  Percentage of subjects who experience 1 or more adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: John N Allan, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WCM Joint Clinical Trials Office — https://jcto.weill.cornell.edu/